CLINICAL TRIAL: NCT05407610
Title: Comparison of Conventional and Cooled Radiofrequency Treatment of the Genicular Nerves Versus Sham Procedure for Patients With Chronic Knee Pain: a Multicentre, Double Blind, Randomised Controlled Trial
Brief Title: Comparison of Conventional and Cooled Radiofrequency of the Genicular Nerves in Patients With Chronic Knee Pain
Acronym: COGENIUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government); Klinische Epidemiologie en Medical Technology Assessment (Unknown)
Responsible Party: Principal Investigator, Jan Van Zundert, Professor, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COGENIUS; Z-2021109 (Other: Ziekenhuis Oost-Limburg); KCE20-1255 (Other Grant/Funding Number: Belgium Health Care Knowledge Centre)
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis; Persistent Postsurgical Pain; Chronic Knee Pain
Keywords: Osteoarthritis; Persistent Postsurgical Pain; Knee; Radiofrequency ablation
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Three-arm, pragmatic, prospective, multicentre, double blind, randomised sham-controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Radiofrequency of the genicular nerves (Active Comparator): In the conventional radiofrequency group a intervention of 80°C at the tip is applied during 90 seconds at each nerve (superolateral, superomedial and inferomedial genicular nerves). The probe stays in place for 150 seconds at each nerve so that the time needed for each procedure is similar.
  Interventions: Procedure: Conventional Radiofrequency ablation of the genicular nerves
- Cooled Radiofrequency of the genicular nerves (Active Comparator): In the cooled radiofrequency group a intervention of 60°C measured at the tip and on average 80°C in the targeted tissue is applied for 150 seconds using the Cooled RF system at each nerve (superolateral, superomedial and inferomedial genicular nerves).
  Interventions: Procedure: Cooled Radiofrequency ablation of the genicular nerves
- Sham procedure (Sham Comparator): In the sham group a 18 gauge introducer and probe will be placed but no RF intervention will be applied. The generator will be turned on without connection to the probe for 150 seconds and the sound of the generator will be mimicked with a recording. The position of the needle will not be checked by fluoroscopy; however, the intervention team will position the fluoroscopy arm and mention the acquisition of the fluoroscopic image to the patient. This way no unnecessary radiation is used.
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Conventional Radiofrequency ablation of the genicular nerves — Conventional Radiofrequency treatment of the genicular nerves of the knee blocks the transmission of painful stimuli from the sensory genicular nerves of the knee to the central nervous system by means of a thermal lesion created using RF current.
  Other Names: Conventional Radiofrequency ablation
  Arms: Conventional Radiofrequency of the genicular nerves
Procedure: Cooled Radiofrequency ablation of the genicular nerves — Cooled RF treatment causes a larger lesion size compared to conventional RF by means of internal cooling of the probe.
  Other Names: Cooled Radiofrequency ablation
  Arms: Cooled Radiofrequency of the genicular nerves
Procedure: Sham procedure — Sham procedure with placing of needles subcutaneously.
  Arms: Sham procedure

SUMMARY:
Chronic knee pain remains a disabling disease despite current treatment strategies. There is an increase in the prevalence of osteoarthritis (OA) of the knee in the general population, presently affecting approximately 450,000 individuals in Belgium. A total knee replacement is a viable alternative for severe knee OA that does not respond to conservative therapy. Unfortunately, up to 53% of patients who undergo a total knee replacement develop persistent post-surgical pain (PPSP). There is currently no effective therapy for PPSP.

A radiofrequency (RF) treatment applies high frequency current on the nerve responsible for pain conduction, resulting in an interruption of the transmission of pain. This can be applied to the nerves innervating the knee joint - the superolateral, superomedial and inferomedial genicular nerves - and could be an alternative, minimally invasive treatment for patients with knee OA who fail conservative treatments and for patients with PPSP. Data from the recent literature indicates that this treatment leads to a reduction of pain intensity and could result in an improvement of knee function, of the psychological state of the individual, and finally in an increase in health-related quality of life. Furthermore, RF of the genicular nerves could help avoid or delay a total knee replacement therefore potentially contributing to cost reduction. Both cooled and conventional RF treatments are reported in the literature to improve pain. The use of water to cool the RF electrodes results in an increased lesion size by removing heat from adjacent tissue, allowing power delivery to be increased. As a consequence, cooled RF could result in a higher chance of success and longer duration of effect. Until now, the studies performed on cooled RF are industry initiated and a direct comparison between conventional, cooled and a sham procedure is lacking.

The aim of the COGENIUS trial is to investigate the effect of the two types of RF treatment on individuals experiencing chronic knee pain that is resistant to conservative treatments. For this purpose, the efficacy and cost-effectiveness of cooled and conventional RF will be compared to a sham procedure in patients suffering from knee OA and PPSP after total knee replacement.

DETAILED DESCRIPTION:
In this three-arm, pragmatic, prospective, multicentre, double blind, randomised sham-controlled trial of approximately 4 years duration, 400 patients with chronic moderate to severe anterior knee pain (>12 months) refractory to conventional treatments will be included. Two groups of chronic knee pain patients will be enrolled depending on the aetiology of knee pain: OA and PPSP. Each patient will undergo a run-in period of 1 to 3 months depending on the previous treatments of the patient. A run-in period is added to the trial to guarantee that conservative treatment is performed in an optimal way before randomisation. In each group (osteoarthritis and persistent post-surgical pain), non-responders to the run-in period will be randomly allocated to a conventional RF intervention of the genicular nerves, a cooled RF intervention of the genicular nerves or a sham procedure in a 2:2:1 ratio. The patients will be followed up for a period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained before any study assessment is performed.
* Adult patients (Age ≥ 18 years old).
* Chronic anterior knee pain (> 12 months) that is moderate to severe (defined as NRS > 4 on most or all days for the index knee either constantly or with motion at time of screening and, an average NRS score reported in the patient diary >4 at the end of the run-in period).
* Unresponsive (meaning insufficient pain reduction or intolerance) to conventional treatments ongoing for at least 12 months prior to inclusion. Conventional treatments must include all of the following: active physiotherapy, pharmacological treatment of pain and intra-articular corticosteroid infiltration.
* Only for patients with Osteoarthritis (OA): Radiologic confirmation of knee osteoarthritis of grade 2 (mild), 3 (moderate) or 4 (severe) noted within 12 months prior to the screening for the index knee according the Kellgren Lawrence criteria diagnosed by an independent radiologist with experience in musculoskeletal imaging on radiography (Rx) or magnetic resonance imaging (MRI). If imaging will need to be performed at screening it is recommended to perform an MRI instead of Rx. Imaging with MRI will enable the independent radiologist to perform a better estimation of the grade of OA.
* Only for patients with Persistent Post-Surgical Pain (PPSP) after Total Knee Arthroplasty (TKA): Patients with PPSP* after TKA need to have had a negative orthopaedic work-up

Exclusion Criteria:

* Local or systemic infection (bacteraemia).
* Evidence of inflammatory arthritis or an inflammatory systemic disease responsible for knee pain.
* Intra-articular injections (steroids, hyaluronic acid, platelet enriched plasma, ...) in the index knee during the 3 months prior to procedure.
* Pregnant, nursing or planning to become pregnant before the study intervention. Participants who become pregnant after the study intervention during the follow-up period will not be excluded.
* Chronic widespread pain.
* Patients with unstable psychosocial disorder.
* Allergies to products used during the procedure (lidocaine, propofol, chlorhexidine).
* Uncontrolled coagulopathy defined as supratherapeutic dose of anticoagulation medication.
* Uncontrolled immune suppression.
* Participating in another clinical trial/investigation within 30 days prior to signing informed consent.
* Patient is currently implanted with a neurostimulator.
* Current radicular pain in index leg.
* Previous conventional or cooled radiofrequency of the index knee.
* Patients with bilateral knee pain defined as chronic knee pain (> 12 months) in both knees that is moderate to severe (defined as a numeric rating scale (NRS) > 4 on most or all days either constantly or with motion) and that is unresponsive (meaning insufficient pain reduction or intolerance) to conventional treatments ongoing for at least 12 months prior to inclusion. Conventional treatments must include all of the following: active physiotherapy, pharmacological treatment of pain and intra-articular corticosteroid infiltration.
* Patients who have a planned TKA in the near future defined as patients who already have agreed on a date for the TKA procedure.
* Patients who are unwilling or mentally incapable to complete the study questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at 6 months post-intervention | 6 months post-intervention.
  The primary endpoint is the WOMAC score (range 0-96) at 6 months post-intervention.
  The WOMAC score is derived from a self-administered osteoarthritis-specific validated questionnaire on pain, stiffness, and physical functioning of the knee joint.The lower the score, the lower the osteoarthritis-specific symptoms are.

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score. | 1-, 3-, 6-, 12- and 24-months post-intervention.
  The WOMAC score (range 0-96) is derived from a self-administered osteoarthritis-specific validated questionnaire on pain, stiffness, and physical functioning of the knee joint.The lower the score, the lower the osteoarthritis-specific symptoms are.
Pain Intentisty | 1-, 3-, 6-, 12- and 24-months post-intervention.
  Pain intensity expressed by the Numerical Rating Scale (NRS) (range 0-10). The NRS score at each visit will be calculated as the mean score of the 4 days prior to each visit.The lower the score, the least pain the patient experiences.
The proportion of patients with a pain reduction of at least 50% compared to baseline expressed by the numerical rating scale (NRS) | 1-, 3-, 6-, 12- and 24-months post-intervention.
  The proportion of patients with a pain reduction of at least 50% compared to baseline expressed by the numerical rating scale (NRS) (0-10). The NRS score at each visit will be calculated as the mean score of the 4 days prior to each visit.The lower the score, the least pain the patient experiences.
Health-related quality of life | 1-, 3-, 6-, 9-, 12- and 24-months post-intervention.
  Health-related quality of life assessed by the EuroQoL-5D-5L (EQ-5D-5L). The questionnaire consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and a visual assessment scale. Responses to the 5 items (one for each dimension) result in a patient's health state that can be transformed into a utility score ranging between 0 (death) and 1 (full health), representing the quality of life of the health state. For the visual assessment scale section, the patient indicates their impression of health on the visual scale. The scale has the following distribution: 0 indicating "worse possible health" and 100 indicating "best possible health".
Goniometry | 1-, 3-, 6-, 12- and 24-months post-intervention.
  Goniometry (maximal knee flexion and extension expressed in degrees) is assessed using the CJOrtho app. The degrees range from 0 to 180 degrees.
'Timed up and Go' test | 1-, 3-, 6-, 12- and 24-months post-intervention.
  The 'Timed up and Go' test assesses the physical functioning of the patient.
The 6-minute walk test | 1-, 3-, 6-, 12- and 24-months post-intervention.
  The 6-minute walk test assesses the physical functioning of the patient. The distance in meters covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
The Hospital Anxiety and Depression Scale (HADS) | 1-, 3-, 6-, 12- and 24-months post- intervention.
  The Hospital Anxiety and Depression Scale (HADS) assesses and detect anxiety and depression in patients with physical health problems. The questionnaire consists of 14 items: 7 items to measure anxiety and 7 items to measure depression.
The Pain Catastrophizing Scale (PCS) | 1-, 3-, 6-, 12- and 24-months post- intervention.
  The Pain Catastrophizing Scale (PCS) assesses the mental health of the patient.The 13 item questionnaire consists of 3 subscales (magnification, rumination and helplessness) and asks patients to reflect on past painful experiences and to indicate the degree on which they experiences each of 13 thoughts of feelings on a 5- point scale (0 not at all and 4 all the time).
Patient Global Impression of Change (PGIC) | 1-, 3-, 6-, 12- and 24-months post- intervention.
  Patients' Patient's Global Impression of Change (PGIC) scale is a self-reported measure that reflects the patient's belief about the treatment efficacy. The patient is asked to rate the efficacy of the treatment on a scale of 1 (much better) to 7 (much worse).
Patient's satisfaction | 1-, 3-, 6-, 12- and 24-months post- intervention.
  Patient's satisfaction assessed by 7-point Likert scale with 0 representing total dissatisfaction and 10 representing maximal satisfaction.
Medication use | 1-, 3-, 6-, 9-, 12- and 24-months post- intervention.
  Medication use measured by Medication Quantification Scale III (MQS III).It computes a single numeric value for a patient's pain medication profile. This number is used to track pain levels through a treatment course or research study.
Opioid dependence | 1-, 3-, 6-, 9-, 12- and 24-months post- intervention.
  The patient is strong opioid dependent if the patient takes an opioid analgesic with the exception of analgesics with tramadol or codeine.
Incidence of related adverse events | Follow-up until 24-months post- intervention.
  The incidence of related adverse events. Active capture during each study contact to assess specific symptoms and adverse events relevant to chronic knee pain or RF intervention.
Health care resource utilisation | Follow-up until 24-months post- intervention.
  The health care resource use questions are created for the COGENIUS study to collect information regarding the visits to a medical specialist (doctor or nurse) or general practitioner as a result of knee pain.
Productivity loss due to sickness | Follow-up until 24-months post- intervention.
  Productivity loss due to sickness assessed by the Work Productivity and Activity Impairment (WPAI). Productivity loss due to sickness refers to output loss resulting from work absence and/or reduced labour input due to sickness. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.

OTHER OUTCOMES:
Phenotype of patients suffering from Persistent Post-Surgical Pain (PPSP) | Baseline
  Demographic data collected at baseline will be used to phenotype patients suffering from PPSP.
Time to additional interventions | Follow-up until 24-months post- intervention.
  Time to additional interventions at each time point. Interventions will be divided in minimally invasive interventions (intraarticular (IA) steroid injections, IA hyaluronic acid, platelet rich plasma of infiltrations, repeat RF of the genicular nerves) and surgery (primary/revision total knee arthroplasty and other knee related surgery) during the follow-up.

CONTACTS AND LOCATIONS:
Locations (15):
- Belgium (13):
  - UZ Antwerpen, Antwerp
  - AZ Klina, Brasschaat
  - ULB Erasme, Brussels
  - UCL Saint-Luc, Brussels
  - Ziekenhuis Oost-Limburg AV, Genk
  - AZ Maria Middelares, Ghent
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHR de la Citadelle, Liège
  - CHU Liège, Liège
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout
- Netherlands (2):
  - Rijnstate, Arnhem
  - MUMC, Maastricht

IPD SHARING:
Plan to Share IPD: Yes
Researcher will need to contact ctu@zol.be in order to request the 'Data Sharing Application' form. Users will need to complete an application form, 'Request for Data Sharing'. The application will be reviewed by the Trial Steering Committee with regard to feasibility and confidentiality. When the application is approved by the Trial Steering Committee, the applicant will be requested to sign a 'Data Use Agreement'. This Data Use Agreement shall be countersigned by ZOL as Sponsor and the CI of the COGENIUS study.
Time Frame: Considering that ongoing research contributing to the completion of datasets must not be compromised by premature or opportunistic sharing and analysis of data, ZOL will not release the data of its studies until the primary study results have been published, unless authorized for release has been granted.

REFERENCES:
- [Derived] Vanneste T, Belba A, van Kuijk S, Kimman M, Bellemans J, Bonhomme V, Sommer M, Emans P, Vankrunkelsven P, Tartaglia K, Van Zundert J. Comparison of conventional and cooled radiofrequency treatment of the genicular nerves versus sham procedure for patients with chronic knee pain: protocol for a multicentre, double-blind, randomised controlled trial (COGENIUS). BMJ Open. 2023 Aug 2;13(8):e073949. doi: 10.1136/bmjopen-2023-073949. PMID 37532482